CLINICAL TRIAL: NCT04536727
Title: Enhancing Well-Being Through Exercise During Old Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, David Xavier Marquez, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013-1027
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2022-10

CONDITIONS: Depression; Osteoarthritis
Keywords: physical activity; exercise; mental health; older adults
MeSH Terms: conditions — Depression; Osteoarthritis; Motor Activity; Psychological Well-Being | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the intervention or wait-list group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The 8-week intervention will consist of the Fit & Strong! program adapted to address the impact of exercise on enhancing positive affect and reducing negative affect and depressive symptoms. Exercise classes will meet three times per week for 90 minutes per session for eight weeks. Each class is divided into 60 minutes of strength training, flexibility, and cardiovascular exercise and 30 minutes of group education/discussion, which has been adapted to include affect-oriented content.
  Interventions: Behavioral: Fit & Strong!
- Wait list (Placebo Comparator): Participants randomized to the wait list group, receive the 8-week Fit & Strong! intervention after the intervention group has completed it.
  Interventions: Behavioral: Wait list

INTERVENTIONS:
Behavioral: Fit & Strong! — The 8-week intervention will consist of the Fit & Strong! program adapted to address the impact of exercise on enhancing positive affect and reducing negative affect and depressive symptoms. Exercise classes will meet three times per week for 90 minutes per session for eight weeks. Each class is divided into 60 minutes of strength training, flexibility, and cardiovascular exercise and 30 minutes of group education/discussion, which has been adapted to include affect-oriented content
  Arms: Intervention
Behavioral: Wait list — Participants randomized to the wait list group receive the 8-week Fit & Strong! intervention after the intervention group has competed it and after the wait list group has provided their post-outcomes.
  Arms: Wait list

SUMMARY:
Determine the feasibility of adapting Fit & Strong!, an evidence-based group physical activity and health education program, to include affect and mood-related content and of employing this intervention among older adults with a range of depressive symptoms.

DETAILED DESCRIPTION:
The specific aims of this pilot are to use a small randomized controlled trial (RCT) with a wait list control design to: 1) Determine the feasibility of adapting Fit & Strong! to include affect and mood-related content and of employing this intervention among older adults with a range of depressive symptoms. 2) Begin to determine whether Fit & Strong! is efficacious as an approach for improving positive affect, reducing negative affect, decreasing symptoms of depression, and improving cognition among older adults. 3) Explore the relationship between negative/positive affect and symptoms of depression and maintenance of physical activity between baseline and 2 months, in order to determine whether improved positive affect and reduced negative affect and depression and improved cognition are associated with an increase in physical activity.

ELIGIBILITY:
Inclusion Criteria:

* ages 60+;
* Sufficient visual and hearing capacity to follow instructions;
* a score of at least 1 on the Patient Health Questionnaire-8 (Kroenke et al., 2001);
* Six Item Screener (Callahan, 2002) score > 4;
* pass screening with the Exercise Assessment and Screening for You (EASY) scale [Cardinal et al., 1996] or have doctor's clearance to participate;
* no recent (<6 months) joint replacements;
* physically inactive (<150 minutes of exercise per week);
* able to walk at least 20 feet (with or without the aid of a cane or walker);
* speak English proficiently.

Exclusion Criteria:

* Non-proficient in English;
* 0 on the Patient Health Questionnaire-8 (Kroenke et al., 2001);
* Six Item Screener < 5 (Callahan, 2005);
* fail screening with the EASY scale and does not have doctor's clearance to participate;
* joint replacement in last 6 months;
* 150+ minutes of exercise per week;
* unable to walk at least 20 feet;
* severe medical illness (i.e., metastatic cancer, brain tumors, unstable cardiac, hepatic, or renal disease, myocardial infarction or stroke) within the 3 months preceding the study;
* Other brain/neurological disorders (i.e., dementia or delirium according to Diagnostic and Statistical Manual (DSM-IV) criteria, history of severe head trauma, Parkinson's disease or Parkinson's plus syndromes, multiple sclerosis, epilepsy);
* Conditions often associated with depression (i.e., endocrinopathies other than diabetes, lymphoma, and pancreatic cancer).

Potential participants for the optional MRI component will be excluded for the following:

* cardiac pacemaker or defibrillator
* metal parts in head, spinal cord, eyes, or chest
* past operation or radiation therapy with skull or brain: e) aneurysm clips
* dentures that have been surgically implanted with magnets, braces:
* claustrophobia:
* heart valve replacement:
* history of work with metal resulting in an injury:
* eye injury with metal:
* history of strokes/seizures:

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Wait List
Started | 13 | 15
Completed | 12 | 13
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Wait List | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.31 (7.36) | 70.27 (9.04) | 69.82 (8.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 15 | 28
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Attendance of the Fit & Strong! Intervention Classes
Description: Total number of Fit & Strong! classes attended (0 to 24 classes).
Time Frame: Baseline, 8 weeks
Population: The Fit & Strong! classes were offered at a residential senior housing development. The wait list classes were scheduled to begin in Winter 2020, however due to Covid, the facility was locked down and classes could not be delivered to the wait list participants.
Measure: Median (Standard Deviation); unit: Classes attended
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 0
Classes attended | 10 (6.94) |

2. Primary Outcome: Acceptability of Fit & Strong! Intervention
Description: Positive evaluation of the intervention assessed during the debriefing session
Time Frame: Baseline, 8 weeks
Population: Anonymous evaluations were given to intervention participants, however the evaluation documents were lost at the site. The site, a senior residential housing complex, was then locked down for Covid and the wait list class was canceled and never held.
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Depressive Symptoms - Emotional Well-being Scale
Description: Assessed by self-administered questionnaire, respondents indicated how much of the time during the past 30 days- "all,""most,""some,""a little,"or "none of the time"-they felt six symptoms of positive affect. The positive affect symptoms are (1) cheerful, (2) in good spirits, (3) extremely happy,(4) calm an peaceful, (5) satisfied, and (6) full of life. Scores ranges from 6-36, with lower a score indicating greater reported emotional well-being. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 1.45 (4.57) | 1.42 (3.58)

4. Secondary Outcome: Physical Activity Scale for the Elderly (PASE)
Description: The PASE score combines information on leisure, household and occupational activity. The PASE assesses the types of activities typically chosen by older adults (walking, recreational activities, exercise, housework, yard work, and caring for others. It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 12.11 (97.92) | -16.86 (46.71)

5. Secondary Outcome: Motor Function - Grip Strength (Dominant Hand)
Description: Participants are seated in a chair with their feet touching the ground. With the elbow bent to 90 degrees and the arm near the trunk, wrist at neutral, participants squeeze the dynamometer as hard as they can for a count of three. The dynamometer provides a digital reading of force in pounds. Greater force (in pounds) represents greater strength. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Pounds | -1.65 (9.51) | -2.39 (14.32)

6. Secondary Outcome: Cerebral Functional Connectivity - Default Mode Network
Description: Functional connectivity is defined as a correlation of the blood oxygenation level dependent (BOLD) signal from each brain network defined by pre-specified regions of interest. Whole-brain images were acquired on a General Electric Magnetic Resonance (GE MR) 750 Discovery 3-T scanner using an 8-channel head coil. Functional connectomes were generated using the resting state functional magnetic resonance imaging (fMRI) toolbox. An increase shows improvement. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Population: Sub-sample of study sample.
Measure: Mean (Standard Deviation); unit: Average functional connectivity
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 4 | 4
Average functional connectivity | .0022 (.2704) | .0921 (.2046)

7. Secondary Outcome: Cerebral Functional Connectivity - Frontoparietal Network
Description: Functional connectivity is defined as a correlation of the blood oxygenation level dependent (BOLD) signal from each brain network defined by prespecified regions of interest. Whole-brain images were acquired on a GE MR 750 Discovery 3-T scanner using an 8-channel head coil. Functional connectomes were generated using the resting state functional magnetic resonance imaging (fMRI) toolbox. An increase shows improvement. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Population: A sub-sample of the study sample.
Measure: Mean (Standard Deviation); unit: Average functional connectivity
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 4 | 4
Average functional connectivity | .0583 (.2128) | .0593 (.3232)

8. Secondary Outcome: Motor Function - Grip Strength (Non-dominant Hand)
Description: as for outcome 5
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Pounds | -5.33 (5.00) | -0.34 (9.51)

9. Secondary Outcome: Motor Function - Peg Board (Dominant Hand)
Description: This simple test of manual dexterity records the time required for the participant to accurately place and remove nine plastic pegs into a plastic pegboard. The 9-Hole Pegboard Dexterity Test provides a score for each hand, with the primary NIH Toolbox score being the number of seconds it takes the participant to complete the task using his/her dominant hand. The raw score is commonly used for interpretation, with faster completion times (less time to complete) representing better manual dexterity. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Time in seconds
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Time in seconds | -1.66 (8.85) | -0.42 (5.56)

10. Secondary Outcome: Gait Speed
Description: Four meter walk test: Participants walk four meters at their usual pace. Participants complete one practice and then two timed trials. Score is the number of seconds it takes to walk four meters, using the better of two trials. A smaller score is better, reflecting faster walking speed. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Time in seconds
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Time in seconds | -1.32 (2.75) | -0.76 (3.96)

11. Secondary Outcome: Cognition - Auditory Verbal Learning (Rey)
Description: The Rey is a word-list learning task in which 15 unrelated words are presented orally (via audio recording) over three consecutive learning trials1. After each presentation, the participant is asked to recall as many of the words as he/she can. The Rey is scored by taking the sum of the number of words recalled across all trials (possible range is 0-45 words). The raw score is most commonly used for interpretation of the Rey test, with higher scores representing better episodic memory. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Words
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Words | -0.5 (2.99) | 3.54 (4.88)

12. Secondary Outcome: Balance - Standing Balance Test
Description: The Standing Balance Test is a measure developed to assess static standing balance. It involves the participant assuming and maintaining up to five poses for 50 seconds each. The sequence of poses is: eyes open on a solid surface, eyes closed on a solid surface, eyes open on a foam surface, eyes closed on a foam surface, eyes open in tandem stance on a solid surface. Postural sway is recorded for each pose using an iPod Touch that the participant wears at waist level. The participant's anterior-posterior postural sway information is fed wirelessly to the iPad. A Fully Corrected T-Score is utilized for the interpretation of normative scores that takes into account gender, age, ethnicity and education differences. Fully Corrected T Scores range from 23 - 77 with higher score indicating better balance. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Score on a scale | -11.56 (10.51) | -2.5 (18.58)

13. Secondary Outcome: Cognition - Dimensional Change Card Sort (DCCS)
Description: DCCS is a measure of cognitive flexibility. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). Scoring is based on a combination of accuracy and reaction time. Scores range from 0 - 45. Higher scores indicate higher levels of cognitive flexibility. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Units on a scale | 1.36 (4.41) | .08 (3.43)

14. Secondary Outcome: Cognition - Flanker Inhibitory Control and Attention
Description: The Flanker task measures both a participant's attention and inhibitory control. The test requires the participant to focus on a given stimulus while inhibiting attention to stimuli flanking it. Sometimes the middle stimulus is pointing in the same direction as the "flankers" (congruent) and sometimes in the opposite direction (incongruent). Scoring is based on a combination of accuracy and reaction time. Scores range from 0 - 45, higher scores indicate higher levels of ability to attend to relevant stimuli and inhibit attention from irrelevant stimuli. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Score on a scale | -0.09 (3.33) | -0.38 (2.81)

15. Secondary Outcome: Cognition - List Sorting
Description: The List Sorting test requires immediate recall and sequencing of different visually and orally presented stimuli (i.e., "working memory"). Pictures of different foods and animals are displayed with accompanying audio recording and written text (e.g., "elephant"), and the participant is asked to say the items back in size order from smallest to largest, first within a single dimension (either animals or foods, called 1-List) and then on two dimensions (foods, then animals, called 2-List). List Sorting is scored by summing the total number of items correctly recalled and sequenced on 1-List and 2-List, which can range from 0-26. Higher scores indicate higher levels of working memory. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Score on a scale | -2.36 (2.66) | 0.31 (2.75)

16. Secondary Outcome: Cognition - Oral Symbol Digit Test
Description: In this test, a coding key with nine abstract symbols is presented - each paired with a number between 1 and 9. Participants are asked to orally indicate which numbers go with symbols that are presented on a sheet of paper. The participant is given 120 seconds to call out as many numbers that go with the corresponding symbols as he/she can - without skipping any. The Oral Symbol Digit Test is scored as the number of items answered correctly in 120 seconds (possible range is 0-144), higher scores representing better processing speed. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Score on a scale | -0.91 (10.77) | 3.58 (9.76)

17. Secondary Outcome: Cognition - Pattern Comparison Processing Speed Test
Description: This test measures speed of processing by asking participants to discern, as quickly as possible, whether two side-by-side pictures are the same or not. The items are presented one pair at a time on the iPad screen, and the participant is given 85 seconds of response time (excluding any time needed for the given iPad to "load" the items) to respond to as many items as possible. Raw scores range from 0-130, higher scores indicate faster speed of processing. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 4.09 (8.89) | 1.92 (7.35)

18. Secondary Outcome: Cognition - Picture Sequence Memory Test
Description: The Picture Sequence Memory Test (PSMT) is a measure developed for the assessment of episodic memory. It involves recalling increasingly lengthy series of illustrated objects and activities that are presented in a particular order on the iPad screen, with corresponding audio-recorded phrases played. The participants are asked to recall the sequence of pictures demonstrated over two learning trials. The PSMT is a measure of episodic memory, which involves the acquisition, storage and effortful recall of new information. Age-corrected normative scores are reported on a scale of 59-140 with with higher scores representing better episodic memory. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 5.44 (11.19) | 5.22 (11.76)

19. Secondary Outcome: Apathy Evaluation Scale (AES) Self
Description: The AES addresses characteristics of goal directed behavior that reflects apathy including behavioral, cognitive, and emotional indicators. Scores range 18-72 (higher scores reflect more apathy). Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 1.0 (4.5) | -.83 (5.24)

20. Secondary Outcome: Balance Confidence Scale
Description: The Balance Confidence Scale is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. Items are rated on a rating scale that ranges from 0 - 100. Score of zero represents no confidence, a score of 100 represents complete confidence. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | -2.15 (12.24) | -6.04 (7.72)

21. Secondary Outcome: Perceived Stress Scale 10-item (PSS-10)
Description: The PSS-10 is a self-reported scale to assess the degree to which one perceives his/her life as stressful. Items are on a 5-point Likert scale ranging from 0 (never) to 4 (very often), indicating how often they have felt or thought a certain way within the past month. Scores range from 0 to 40, higher scores indicate greater perceived stress. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 2.45 (6.04) | 1.46 (4.54)

22. Secondary Outcome: Satisfaction With Life Scale
Description: A 5-item scale designed to measure global cognitive judgments of one's life satisfaction (not a measure of either positive or negative affect). Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. Scores range from 5 to 35 with a higher score indicating greater satisfaction with life. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | -2.00 (5.08) | 0.23 (4.68)

23. Secondary Outcome: Self-Efficacy for Exercise
Description: Adapted from the Chronic Disease Self-Efficacy Scales, this scale assesses the participants confidence safely performing different types of exercise. The scale consists of 4 items rated on a scale from 1 (least confidence) to (most confidence). Scale score range is 1-10, with a higher score indicated greater confidence. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 0.23 (1.63) | 0.00 (1.68)

24. Secondary Outcome: Snaith-Hamilton Pleasure Scale (SHAPS)
Description: The SHAPS is a 14-item scale that measures anhedonia, the inability to experience pleasure. Responses range from 0 Strongly Agree to 3 Strongly Disagree. Scores range from 0 - 42, with higher score indicating greater anhedonia. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 2.00 (5.92) | 0.45 (4.01)

25. Secondary Outcome: Timed Up and Go (TUG)
Description: The TUG is an assessment of mobility, balance, walking ability, and fall risk in older adults. Participants are instructed to stand up from a chair, walk 3 meters at a comfortable pace, walk back to the chair and sit down. The score is the time in seconds to perform the task. A lower score indicates better ability. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
Seconds | 0.43 (4.38) | 0.19 (2.53)

26. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: The WOMAC is a self-reported assessment of osteoarthritis symptoms in the lower body. Questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Total WOMAC score ranges from 0-96, with a higher score indicating greater osteoarthritis symptomatology. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | 8.00 (14.95) | 5.91 (12.17)

27. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Scores range from 0-30 with a higher score meaning better cognitive function. Change from baseline to post-test follow-up at 8-weeks is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Wait List
Number analyzed (Participants) | 13 | 15
score on a scale | -1.91 (3.36) | -1.4 (3.27)

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Intervention | Wait List
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT04536727/Prot_SAP_000.pdf